CLINICAL TRIAL: NCT00691028
Title: Clinical Study to Assess the Efficacy and Safety of Increased Dose of TA-650(Infliximab) in Patients With Rheumatoid Arthritis
Brief Title: Efficacy and Safety of Increased Dose of TA-650(Infliximab) in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: General Manager, Clinical Research Department III, Mitsubishi Tanabe Pharma Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-650-13; JapicCTI-050146
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; Infliximab; TA-650; Remicade
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TA-650 3 mg/kg (Experimental)
  Interventions: Drug: TA-650 3 mg/kg
- TA-650 6 mg/kg (Experimental)
  Interventions: Drug: TA-650 6 mg/kg
- TA-650 10 mg/kg (Experimental)
  Interventions: Drug: TA-650 10 mg/kg

INTERVENTIONS:
Drug: TA-650 3 mg/kg — 3 mg/kg of TA-650 will be intravenously infused over a period of more than 2 hours at weeks 0, 2 and 6. Then 3 mg/kg of TA-650 will be intravenously infused over a period of more than 2 hours at weeks 14, 22, 30, 38 and 46.
  Other Names: Infliximab; REMICADE
  Arms: TA-650 3 mg/kg
Drug: TA-650 6 mg/kg — 3 mg/kg of TA-650 will be intravenously infused over a period of more than 2 hours at weeks 0, 2 and 6 weeks. Then 6 mg/kg of TA-650 will be intravenously infused over a period of more than 2 hours at weeks 14, 22, 30, 38 and 46.
  Other Names: Infliximab; REMICADE
  Arms: TA-650 6 mg/kg
Drug: TA-650 10 mg/kg — 3 mg/kg of TA-650 will be intravenously infused over a period of more than 2 hours at weeks 0, 2 and 6. Then 10 mg/kg of TA-650 will be intravenously infused over a period of more than 2 hours at weeks 14, 22, 30, 38 and 46.
  Other Names: Infliximab; REMICADE
  Arms: TA-650 10 mg/kg

SUMMARY:
The purpose of this study is to assess the efficacy, safety and pharmacokinetics of maintenance treatment with 3mg/kg, 6mg/kg or 10mg/kg of TA-650 in combination with methotrexate (MTX) after three infusions (weeks-0, 2, 6) of 3mg/kg in Rheumatoid Arthritis (RA) showing an insufficient response to MTX.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active RA in spite of stable dose of MTX

Exclusion Criteria:

* Having received infliximab in the past
* Having a history of serious infection which caused hospitalization within 6 months before the registration
* Having an active tuberculosis
* Having a complication or a history of malignancy within 5 years before the registration

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2005-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

REFERENCES:
- [Background] Takeuchi T, Miyasaka N, Inoue K, Abe T, Koike T; RISING study. Impact of trough serum level on radiographic and clinical response to infliximab plus methotrexate in patients with rheumatoid arthritis: results from the RISING study. Mod Rheumatol. 2009;19(5):478-87. doi: 10.1007/s10165-009-0195-8. Epub 2009 Jul 22. PMID 19626391
- [Derived] Takeuchi T, Miyasaka N, Inui T, Yano T, Yoshinari T, Abe T, Koike T. High titers of both rheumatoid factor and anti-CCP antibodies at baseline in patients with rheumatoid arthritis are associated with increased circulating baseline TNF level, low drug levels, and reduced clinical responses: a post hoc analysis of the RISING study. Arthritis Res Ther. 2017 Sep 2;19(1):194. doi: 10.1186/s13075-017-1401-2. PMID 28865493

RESULTS

PARTICIPANT FLOW:
Groups:
- TA-650 3 mg/kg: 99 patients received TA-650 at 3mg/kg treatment during the double-blind period starting from week14.
- TA-650 6 mg/kg: 104 patients received TA-650 at 6mg/kg treatment during the double-blind period starting from week14.
- TA-650 10 mg/kg: 104 patients received TA-650 at 10mg/kg treatment during the double-blind period starting from week14.
- Open-label: 327 patients received TA-650 at 3 mg/kg treatment during the open-label period.
Period: Open-label Period
Arm/Group | TA-650 3 mg/kg | TA-650 6 mg/kg | TA-650 10 mg/kg | Open-label
Started | 0 | 0 | 0 | 327
Completed | 0 | 0 | 0 | 307
Not Completed | 0 | 0 | 0 | 20
Not completed — Adverse Event | 0 | 0 | 0 | 16
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3
Not completed — not come to a hospital | 0 | 0 | 0 | 1
Period: Double-blind Period
Arm/Group | TA-650 3 mg/kg | TA-650 6 mg/kg | TA-650 10 mg/kg | Open-label
Started | 99 | 104 | 104 | 0
Completed | 86 | 91 | 95 | 0
Not Completed | 13 | 13 | 9 | 0
Not completed — Adverse Event | 8 | 9 | 6 | 0
Not completed — Lack of Efficacy | 4 | 3 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — not come to a hospital. | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TA-650 3 mg/kg | TA-650 6 mg/kg | TA-650 10 mg/kg | Total
Number analyzed (Participants) | 99 | 104 | 104 | 307
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 89 | 96 | 92 | 277
  >=65 years | 10 | 8 | 12 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (11.7) | 48.8 (11.8) | 50.4 (12.5) | 49.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 86 | 89 | 253
  Male | 21 | 18 | 15 | 54

OUTCOME MEASURES:

1. Primary Outcome: Numeric Index of American College of Rheumatology Response (ACR-N, N Shows the Percent Improvement)
Description: The ACR-N index of improvement is the minimum of the following: (1) the percent decrease from baseline in tender joint counts(TJC) or (2) the percent decrease from baseline in swollen joint counts(SJC) or (3) the median percent decrease from baseline for the following: a. Patient's assessment of pain (visual analog scale (VAS) 0-100, 100 worst pain); b. Patient's global assessment of disease activity (VAS 0-100); c. Physician's global assessment of disease activity (VAS 0-100); d. Physical function as measured by the Health Assessment Questionnaire(HAQ)(0-3); e. C-Reactive Protein(CRP) measurement. Higher numbers (maximum:100) indicate more improvement.
Time Frame: baseline and week 54
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TA-650 3 mg/kg | TA-650 6 mg/kg | TA-650 10 mg/kg
Number analyzed (Participants) | 99 | 104 | 104
percent change | 51.3 (32.1) | 53.8 (34.4) | 58.3 (31.3)

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20, 50 and 70% Response (ACR20, 50, 70)
Description: ACR 20 (50 or 70) response is a decrease of at least 20% (50% or 70%) in both TJC and SJC and in 3 to 5 assessments (patient's assessment of pain [VAS] with 0, no pain to 100, worst pain; patient's and physician's global assessment of disease activity VAS scales: overall disease activity [0, very well to 100, very poor and 0, no arthritis activity to 100, extremely active, respectively]; [HAQ]: 20-questions on life activities [0, no difficulty to 3, inability to perform a task]; [CRP])
Time Frame: 54 weeks
Measure: Number; unit: percentage of participants
Arm/Group | TA-650 3 mg/kg | TA-650 6 mg/kg | TA-650 10 mg/kg
Number analyzed (Participants) | 99 | 104 | 104
percentage of participants
  ACR20% improvement(percentage) | 75.8 | 78.8 | 82.7
  ACR50% improvement (percentage) | 60.6 | 58.7 | 66.3
  ACR70% improvement (percentage) | 37.4 | 42.3 | 43.3

3. Secondary Outcome: Tender Joint Counts (TJC)
Description: The TJC was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The TJC was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1.
Time Frame: 54 weeks
Measure: Mean (Standard Deviation); unit: count
Arm/Group | TA-650 3 mg/kg | TA-650 6 mg/kg | TA-650 10 mg/kg
Number analyzed (Participants) | 99 | 104 | 104
count
  Tender joint count, baseline | 18.6 (11.3) | 18.0 (10.5) | 17.5 (10.9)
  Tender joint count, week54 | 6.3 (8.6) | 4.8 (7.7) | 4.8 (7.6)

4. Secondary Outcome: Swollen Joint Count (SJC)
Description: The SJC was determined by examination of 66 joints and identifying when swelling was present. The SJC was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1.
Time Frame: 54 weeks
Measure: Mean (Standard Deviation); unit: count
Arm/Group | TA-650 3 mg/kg | TA-650 6 mg/kg | TA-650 10 mg/kg
Number analyzed (Participants) | 99 | 104 | 104
count
  Swollen joint count, baseline | 14.2 (6.1) | 13.1 (8.4) | 13.7 (7.3)
  Swollen joint count, week 54 | 3.6 (4.8) | 3.3 (4.6) | 3.0 (4.6)

5. Secondary Outcome: CRP Level
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation. Normal range of CRP is 0 mg/dL to 0.3 mg/dL. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: 54 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | TA-650 3 mg/kg | TA-650 6 mg/kg | TA-650 10 mg/kg
Number analyzed (Participants) | 99 | 104 | 104
mg/dl
  CRP level, baseline | 2.5 [1.3 to 4.1] | 2.3 [1.3 to 3.5] | 2.3 [1.1 to 4.5]
  CRP level, week 54 | 0.5 [0.1 to 2.3] | 0.4 [0.1 to 1.1] | 0.2 [0.1 to 1.0]

6. Secondary Outcome: Change From Baseline in DAS28
Description: DAS28 is calculated using TJC, SJC erythrocyte sedimentation rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x log (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity. A negative change score indicates improvement. Total score range:0 to 9.4, higher score indicated more disease activity. DAS28 =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate disease activity, >5.1 to 9.4 implied high disease activity and <2.6 implied remission.
Time Frame: baseline and week 54
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TA-650 3 mg/kg | TA-650 6 mg/kg | TA-650 10 mg/kg
Number analyzed (Participants) | 99 | 104 | 104
units on a scale | -2.30 (1.56) | -2.57 (1.69) | -2.80 (1.58)

7. Secondary Outcome: Change From Baseline to Week 54 in HAQ
Description: HAQ: patient's assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: 54 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TA-650 3 mg/kg | TA-650 6 mg/kg | TA-650 10 mg/kg
Number analyzed (Participants) | 99 | 104 | 104
units on a scale | -0.48 (0.70) | -0.56 (0.64) | -0.59 (0.63)

8. Secondary Outcome: Change in Modified Total Sharp Score (mTSS) at week54 From Baseline
Description: The mTSS is a measure of change in joint health. Digitized images of radiographs of hands and feet obtained at screening and Week 54 were scored in a blinded manner. Joints were scored for erosions on a scale of 0 (no damage) to 5 and joint space narrowing on a scale of 0 (no damage) to 4. Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 390 [maximal disease]). An increase in mTSS from baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: baseline and week 54
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | TA-650 3 mg/kg | TA-650 6 mg/kg | TA-650 10 mg/kg
Number analyzed (Participants) | 99 | 104 | 104
score | 0.00 [-1.00 to 1.00] | 0.48 [-0.50 to 1.64] | 0.00 [-1.00 to 0.81]

9. Secondary Outcome: Pharmacokinetics- Serum Concentration of Infliximab
Description: Serum level of infliximab was measured by enzyme-linked immunosorbent assay (ELISA), using a monoclonal antibody against infliximab. The lowest level of infliximab that could be reliably detected was 0.1 ug/ml.
Time Frame: 54 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Pharmacokinetics Positive- ATI
Description: ATI (antibody to Infliximab) was measured by a modification of an enzyme immunoassay.
Time Frame: 54 weeks
Measure: Number; unit: participants
Arm/Group | TA-650 3 mg/kg | TA-650 6 mg/kg | TA-650 10 mg/kg
Number analyzed (Participants) | 99 | 104 | 104
participants | 27 | 24 | 13

ADVERSE EVENTS:
Time Frame: 54 weeks
Groups:
- TA-650 3 mg/kg (Double-blind): 99 patients received TA-650 at 3mg/kg treatment during the double-blind period starting from week14.
- TA-650 6 mg/kg (Double-blind): 104 patients received TA-650 at 6mg/kg treatment during the double-blind period starting from week14.
- TA-650 10 mg/kg (Double-blind): 104 patients received TA-650 at 10mg/kg treatment during the double-blind period starting from week14.
Arm/Group | TA-650 3 mg/kg (Double-blind) | TA-650 6 mg/kg (Double-blind) | TA-650 10 mg/kg (Double-blind) | Open-label
Serious Adverse Events (participants affected / at risk) | 7/99 | 5/104 | 9/104 | 17/327
Other Adverse Events (participants affected / at risk) | 93/99 | 93/104 | 96/104 | 153/327
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-650 3 mg/kg (Double-blind) (N=99) | TA-650 6 mg/kg (Double-blind) (N=104) | TA-650 10 mg/kg (Double-blind) (N=104) | Open-label (N=327)
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cryptococcosis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 2
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 2 | 2
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
Anaphylactoid reaction (Immune system disorders) | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TA-650 3 mg/kg (Double-blind) (N=99) | TA-650 6 mg/kg (Double-blind) (N=104) | TA-650 10 mg/kg (Double-blind) (N=104) | Open-label (N=327)
Palpitations (Cardiac disorders) | 0 | 5 | 0 | 7
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 3 | 0
Conjunctivitis (Eye disorders) | 3 | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 5 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 1 | 0
Dental caries (Gastrointestinal disorders) | 2 | 2 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 4 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 3 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 1 | 4 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 2 | 5 | 0
Chest discomfort (General disorders) | 0 | 1 | 3 | 0
Chest pain (General disorders) | 0 | 3 | 2 | 0
Malaise (General disorders) | 0 | 2 | 3 | 0
Pyrexia (General disorders) | 6 | 6 | 4 | 12
Hepatic function abnormal (Hepatobiliary disorders) | 8 | 3 | 3 | 11
Bronchitis (Infections and infestations) | 2 | 5 | 4 | 0
Gastroenteritis (Infections and infestations) | 3 | 2 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 4 | 0
Nasopharyngitis (Infections and infestations) | 29 | 29 | 30 | 56
Oral candidiasis (Infections and infestations) | 2 | 0 | 0 | 0
Paronychia (Infections and infestations) | 4 | 1 | 4 | 0
Pharyngitis (Infections and infestations) | 4 | 0 | 4 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 4 | 0 | 1 | 0
Tinea infection (Infections and infestations) | 1 | 3 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 4 | 0
Alanine aminotransferase increased (Investigations) | 1 | 12 | 14 | 33
Aspartate aminotransferase increased (Investigations) | 1 | 8 | 8 | 20
Blood pressure increased (Investigations) | 1 | 3 | 4 | 11
Gamma-glutamyltransferase increased (Investigations) | 2 | 3 | 1 | 0
Blood urine present (Investigations) | 3 | 4 | 5 | 0
Heart rate increased (Investigations) | 0 | 3 | 0 | 0
Liver function test abnormal (Investigations) | 4 | 3 | 0 | 7
White blood cell count decreased (Investigations) | 1 | 2 | 3 | 0
White blood cell count increased (Investigations) | 3 | 2 | 2 | 0
Protein urine present (Investigations) | 1 | 3 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 4 | 0 | 0
Antinuclear antibody positive (Investigations) | 25 | 15 | 17 | 0
DNA antibody positive (Investigations) | 65 | 58 | 54 | 16
Cell marker increased (Investigations) | 2 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 4 | 4 | 7
Headache (Nervous system disorders) | 8 | 4 | 4 | 7
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 9 | 13
Acne (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 4 | 3 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4 | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 12 | 9 | 18
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 5 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other